CLINICAL TRIAL: NCT03711136
Title: Comparison of Standard and Hybrid Techniques in Surgical Treatment of Proximal Aortic Dissection
Brief Title: Comparison of stAndard and Hybrid Surgical Techniques in the Treatment of proximaL Aortic dissEctions
Acronym: CASTLE
Status: Completed | Type: Observational
Sponsor: Novosibirsk Scientific Research Institute for Circulatory Pathology (Other)
Responsible Party: Principal Investigator, Alexander Edemskiy, cardiovascular surgeon, Novosibirsk Scientific Research Institute for Circulatory Pathology
Other Study IDs: CASTLE
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: State of Non-operated Aortic Segments; Aorto-related Events

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frozen elephant trunk surgery
  Interventions: Procedure: aortic prosthesis
- Standart surgery
  Interventions: Procedure: aortic prosthesis

INTERVENTIONS:
Procedure: aortic prosthesis — ascending aortic and/or aortic arch prosthesis with linear vascular prosthesis or hybrid prosthesis

SUMMARY:
The study is devoted to the evaluation of the results of surgical treatment of patients with proximal aortic dissection. Two groups of patients with standard and hybrid surgery are compared. Early and long-term postoperative results are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* aortic dissection type A

Exclusion Criteria:

* age limits

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with proximal aortic dissection operated using one of the techniques
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Aorto-related events | 3 years
  Death, reoperations,thoracoabdomminal aneurysms

CONTACTS AND LOCATIONS:
Locations (1):
- NRICP, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No